CLINICAL TRIAL: NCT03305419
Title: A Single-centre, Randomized, Double-blind (Sponsor-unblinded), Placebo-controlled Study to Evaluate the Safety, Tolerability and Pharmacokinetics of GSK2982772 in Repeat Oral Doses in Healthy Subjects
Brief Title: A Safety and Pharmacokinetic (PK) Study of GSK2982772 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 205184; 2017-002662-45 (EudraCT Number)
Record Dates: First submitted 2017-10-04; First posted 2017-10-10 (Actual); Results first posted 2019-11-01 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-09

CONDITIONS: Autoimmune Diseases
Keywords: Crossover; Sequential; GSK2982772; Safety; Pharmacokinetics; Healthy subjects
MeSH Terms: conditions — Autoimmune Diseases | interventions — GSK2982772

STUDY DESIGN:
Intervention Model Description: This study will consist of two parts; Part A and Part B. Part A will be a 3-way crossover design and Part B will be a sequential-group design.
Who Masked: Participant, Investigator
Masking Description: This will be a double-blind study. Subjects and investigator will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- Subjects receiving treatment sequence ABC in cohort 1: Part A (Experimental): Eligible subjects will be randomized to receive treatment sequence ABC in Part A; A= GSK2982772 120 mg TID, B= GSK2982772 240 mg TID, and C= GSK2982772 360 mg BID. Subjects will receive oral capsule of GSK2982772 or placebo on Day 1 in each of the 3 treatment periods followed by a wash-out period of at least 7 days between dosing regimens.
  Interventions: Drug: GSK2982772 capsule; Drug: Placebo capsule
- Subjects receiving treatment sequence ABP in cohort 1: Part A (Experimental): Eligible subjects will be randomized to receive treatment sequence ABP in Part A; A= GSK2982772 120 mg TID, B= GSK2982772 240 mg TID, and P= Placebo. Subjects will receive oral capsule of GSK2982772 or placebo on Day 1 in each of the 3 treatment periods followed by a wash-out period of at least 7 days between dosing regimens.
  Interventions: Drug: GSK2982772 capsule; Drug: Placebo capsule
- Subjects receiving treatment sequence APC in cohort 1: Part A (Experimental): Eligible subjects will be randomized to receive treatment sequence APC in Part A; A= GSK2982772 120 mg TID, P= Placebo and C= GSK2982772 360 mg BID. Subjects will receive oral capsule of GSK2982772 or placebo on Day 1 in each of the 3 treatment periods followed by a wash-out period of at least 7 days between dosing regimens.
  Interventions: Drug: GSK2982772 capsule; Drug: Placebo capsule
- Subjects receiving treatment sequence PBC in cohort 1: Part A (Experimental): Eligible subjects will be randomized to receive treatment sequence PBC in Part A; P= Placebo, B= GSK2982772 240 mg TID and C= GSK2982772 360 mg BID. Subjects will receive oral capsule of GSK2982772 or placebo on Day 1 in each of the 3 treatment periods followed by a wash-out period of at least 7 days between dosing regimens.
  Interventions: Drug: GSK2982772 capsule; Drug: Placebo capsule
- Subjects receiving GSK2982772 120 mg TID in cohort 2 : Part B (Experimental): Eligible subjects will receive GSK2982772 oral capsule with a dose of 120 mg TID for 14 days in Part B.
  Interventions: Drug: GSK2982772 capsule
- Subjects receiving GSK2982772 120 mg TID in cohort 3 : Part B (Experimental): Eligible subjects will receive GSK2982772 oral capsule with a dose of 120 mg TID for 14 days in Part B.
  Interventions: Drug: GSK2982772 capsule
- Subjects receiving GSK2982772 240 mg TID in cohort 4: Part B (Experimental): Eligible subjects will receive GSK2982772 oral capsule with a dose of 240 mg TID for 14 days in Part B.
  Interventions: Drug: GSK2982772 capsule
- Subjects receiving GSK2982772 360 mg BID in cohort 5: Part B (Experimental): Eligible subjects will receive GSK2982772 oral capsule with a dose of 360 mg BID for 14 days in Part B.
  Interventions: Drug: GSK2982772 capsule
- Subjects receiving placebo in cohort 2 : Part B (Placebo Comparator): Subjects will receive placebo oral capsule for 14 days in Part B.
  Interventions: Drug: Placebo capsule
- Subjects receiving placebo in cohort 3 : Part B (Placebo Comparator): Subjects will receive placebo oral capsule for 14 days in Part B.
  Interventions: Drug: Placebo capsule
- Subjects receiving placebo in cohort 4 : Part B (Placebo Comparator): Subjects will receive placebo oral capsule for 14 days in Part B.
  Interventions: Drug: Placebo capsule
- Subjects receiving placebo in cohort 5: Part B (Placebo Comparator): Subjects will receive placebo oral capsule for 14 days in Part B.
  Interventions: Drug: Placebo capsule

INTERVENTIONS:
Drug: GSK2982772 capsule — GSK2982772 will be available as size 00, white, opaque capsule containing white to almost white Solid (120 mg maximum fill per capsule). It will be administered orally with water to receive total dose of 120 mg, 240 mg or 360 mg per randomization.
  Arms: Subjects receiving GSK2982772 120 mg TID in cohort 2 : Part B; Subjects receiving GSK2982772 120 mg TID in cohort 3 : Part B; Subjects receiving GSK2982772 240 mg TID in cohort 4: Part B; Subjects receiving GSK2982772 360 mg BID in cohort 5: Part B; Subjects receiving treatment sequence ABC in cohort 1: Part A; Subjects receiving treatment sequence ABP in cohort 1: Part A; Subjects receiving treatment sequence APC in cohort 1: Part A; Subjects receiving treatment sequence PBC in cohort 1: Part A
Drug: Placebo capsule — Placebo will be available as size 00, white, opaque capsule containing white to almost white Solid. It will be administered orally with water.
  Arms: Subjects receiving placebo in cohort 2 : Part B; Subjects receiving placebo in cohort 3 : Part B; Subjects receiving placebo in cohort 4 : Part B; Subjects receiving placebo in cohort 5: Part B; Subjects receiving treatment sequence ABC in cohort 1: Part A; Subjects receiving treatment sequence ABP in cohort 1: Part A; Subjects receiving treatment sequence APC in cohort 1: Part A; Subjects receiving treatment sequence PBC in cohort 1: Part A

SUMMARY:
This study is designed to evaluate the safety, tolerability and PK of GSK2982772, in repeat oral doses in healthy subjects. This study is being conducted to support administration of higher dose levels of GSK2982772 than initially studied in the First Time in Human (FTiH) study. This study will also assess the impact of food during the repeat doses of GSK2982772. This will be a two part study; Part A and Part B. Part A (cohort 1) - single ascending dose, randomized, placebo-controlled, 3-way crossover. Part B (cohorts 2, 3, 4 and 5) - repeat dose, randomized, placebo-controlled, sequential-group. Subjects will be randomized in 3:1 ratio to receive GSK2982772 or placebo in crossover manner on Day 1 of each of the three periods in Part A. Subjects will be randomized in 3:1 ratio to receive GSK2982772 or placebo in sequential groups for 14 days in cohort 2 of Part B and in 9:5 ratio to receive GSK2982772 or placebo in sequential groups for 14 days in cohorts 3, 4 and 5 of Part B. Approximately 66 subjects will be included in this study. The study duration, including screening and follow-up, will not be expected to exceed 13 weeks for Part A and 8 weeks for Part B.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 18 to 65 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by the Investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, neurological examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the Investigator in consultation with the Medical Monitor (if required) agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body weight >=50 kilograms (kg) and body mass index (BMI) within the range 19 - 30 kg per square meter (kg/m^2) (inclusive).
* A male subject with a female partner of reproductive potential must agree to use contraception during the treatment period and for at least 90 days after the last dose of study treatment and refrain from donating sperm during this period. A female subject is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies: not a woman of childbearing potential (WOCBP) or a WOCBP who agrees to follow the contraceptive guidance for a minimum of 28 days prior to the treatment period and for at least 30 days after the last administration of study drug. A WOCBP using a hormonal method of highly effective contraception must also agree to partner use of a male condom during the treatment period and for at least 30 days after the last administration of study drug.
* Capable of giving signed informed consent.

Exclusion Criteria:

* History or presence of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study treatment; or interfering with the interpretation of data.
* History of herpes zoster (shingles) reactivation.
* Evidence of active or latent tuberculosis (TB) as documented by medical history and examination, chest x-rays (posterior anterior and lateral), and TB testing: either a positive tuberculin skin test (TST; defined as a skin induration >5 millimeter (mm) at 48 to 72 hours, regardless of Bacillus Calmette-Guerin (BCG) or other vaccination history) or a positive (not indeterminate) QuantiFERON-TB Gold test.
* ALT >1.5 times upper limit of normal (ULN).
* Bilirubin >1.5 times ULN (isolated bilirubin >1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* ECG QT interval corrected for heart rate (QTc) >450 millisecond (msec).
* History of serious or recurrent infections or has had an active infection within 14 days of receiving study medication.
* History of diagnosis of obstructive sleep apnoea or significant respiratory disorder. Childhood asthma that has fully resolved is permitted.
* Part A: History of active suicidal ideation behavior (SIB) within the past 6 months or any history of attempted suicide in a subject's lifetime.
* History of current evidence of febrile seizures, epilepsy, convulsions, significant head injury, or other significant neurologic conditions.
* Past or intended use of over-the-counter or prescription medication, including herbal medications, within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is the longest) prior to dosing.
* Subject received a vaccine (either live attenuated or now-live) within 30 days prior to randomization, or plans to receive a live attenuated vaccine within 30 days + 5 half-lives (32 days) of the last dose of study medication.
* Participation in the study would result in loss of blood or blood products in excess of 500 milliliters (mL) within a 56-day period.
* Exposure to more than 4 new chemical entities within 12 months prior to the first dosing day.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Presence of Hepatitis B surface antigen (HBsAg) at screening Positive Hepatitis C antibody test result at screening.
* Positive pre-study drug/alcohol screen.
* Positive human immunodeficiency virus (HIV1 and 2) antibody test.
* Regular use of known drugs of abuse.
* Subjects with impaired renal function defined as Chronic Kidney Disease Epidemiology Collaboration (CKS-EPI) Creatinine > 1.6 mg/deciliter (mg/dL) with an age appropriate glomerular filtration rate (GFR) <= 60 (mL/minute/1.73 m^2) estimated by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation.
* An elevated C-reactive protein (CRP) outside of the normal reference range.
* Regular alcohol consumption within 6 months prior to the study defined as: For United Kingdom (UK) - an average weekly intake of >14 units for males and females. One unit is equivalent to 8 grams (g) of alcohol: a half-pint (approximately 240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* Cotinine or carbon monoxide levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Sensitivity to any of the study treatments, or components thereof, or drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates participation in the study.
* Unwilling or unable to swallow multiple size 00 capsules as part of study participation.

PART B Specific exclusion criteria:

* History of SIB as measured using the Columbia Suicide Severity Rating Scale (C-SSRS) or a history of attempted suicide.
* A positive anti-nuclear antibody (ANA) outside of the normal reference range.
* Fasting total cholesterol >=300 mg/dL or triglycerides >=250 mg/dL.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2018-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD is made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency

REFERENCES:
- [Derived] Tompson DJ, Davies C, Scott NE, Cannons EP, Kostapanos M, Gross AS, Powell M, Ino H, Shimamura R, Ogura H, Nagakubo T, Igarashi H, Nakano A. Comparison of the Pharmacokinetics of RIPK1 Inhibitor GSK2982772 in Healthy Western and Japanese Subjects. Eur J Drug Metab Pharmacokinet. 2021 Jan;46(1):71-83. doi: 10.1007/s13318-020-00652-2. PMID 33165774

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study consisted of two parts; part A was single ascending dose, 3-way crossover and part B was repeat dose, sequential assignment which investigated the safety, tolerability, and pharmacokinetics of GSK2982772, in healthy participants.
Pre-assignment Details: A total of 62 participants (15 in Part A and 47 in Part B) were enrolled in the study. Participants were not enrolled into the GSK2982772 360 milligram (mg) twice daily (BID) arm of Part B as one participant in the 360 mg BID dose level in Part A exceeded the maximum concentration (Cmax) stopping criteria.
Groups:
- Part A:GSK2982772 120 mg TID/240 mg TID/360 mg BID: Participants received oral capsule of 120 mg GSK2982772 TID in treatment period 1 followed by 240 mg TID in treatment period 2 followed by 360 mg BID in treatment period 3. The treatment periods were separated by a washout period of at least 7 days.
- Part A:GSK2982772 120 mg TID/240 mg TID/Placebo: Participants received oral capsule of 120 mg GSK2982772 TID in treatment period 1 followed by 240 mg TID in treatment period 2 followed by matching Placebo in treatment period 3. The treatment periods were separated by a washout period of at least 7 days.
- Part A:GSK2982772 120 mg TID/Placebo/GSK2982772 360 mg BID: Participants received oral capsule of 120 mg GSK2982772 TID in treatment period 1 followed by matching Placebo in treatment period 2 followed by 360 mg GSK2982772 BID in treatment period 3. The treatment periods were separated by a washout period of at least 7 days.
- Part A:Placebo/GSK2982772 240 mg TID/360 mg BID: Participants received oral capsule of matching Placebo in treatment period 1 followed by 240 mg GSK2982772 TID in treatment period 2 followed by 360 mg GSK2982772 BID in treatment period 3. The treatment periods were separated by a washout period of at least 7 days.
- Part B:Placebo: Participants received matching oral placebo capsule to GSK2928772 for 14 days.
- Part B:GSK2982772 120 mg TID: Participants received GSK2982772 oral capsule at a dose of 120 mg TID for 14 days
- Part B:GSK2982772 240 mg TID: Participants received GSK2982772 oral capsule at a dose of 240 mg TID for 14 days.
- Part B:GSK2982772 360 mg BID: Participants were planned to receive GSK2982772 oral capsule at a dose of 360 mg BID for 14 days.
Period: Part A Period 1 (1Day) + Washout (7days)
Arm/Group | Part A:GSK2982772 120 mg TID/240 mg TID/360 mg BID | Part A:GSK2982772 120 mg TID/240 mg TID/Placebo | Part A:GSK2982772 120 mg TID/Placebo/GSK2982772 360 mg BID | Part A:Placebo/GSK2982772 240 mg TID/360 mg BID | Part B:Placebo | Part B:GSK2982772 120 mg TID | Part B:GSK2982772 240 mg TID | Part B:GSK2982772 360 mg BID
Started (Par. discontinuation was only collected at FU visits.Thus, treatment & washout periods are combined) | 3 | 3 | 3 | 3 | 0 | 0 | 0 | 0
Completed (Par. discontinuation was only collected at FU visits.Thus, treatment & washout periods are combined) | 3 | 2 | 3 | 3 | 0 | 0 | 0 | 0
Not Completed | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A Period 2 (1Day) + Washout (7days)
Arm/Group | Part A:GSK2982772 120 mg TID/240 mg TID/360 mg BID | Part A:GSK2982772 120 mg TID/240 mg TID/Placebo | Part A:GSK2982772 120 mg TID/Placebo/GSK2982772 360 mg BID | Part A:Placebo/GSK2982772 240 mg TID/360 mg BID | Part B:Placebo | Part B:GSK2982772 120 mg TID | Part B:GSK2982772 240 mg TID | Part B:GSK2982772 360 mg BID
Started (Par. discontinuation was only collected at FU visits.Thus, treatment & washout periods are combined) | 3 | 3 (1 participant was added to GSK2982772 120 mg TID/240 mg TID/Placebo arm) | 3 | 3 | 0 | 0 | 0 | 0
Completed (Par. discontinuation was only collected at FU visits.Thus, treatment & washout periods are combined) | 1 | 3 | 3 | 3 | 0 | 0 | 0 | 0
Not Completed | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A Period 3 (1Day) + Washout (7days)
Arm/Group | Part A:GSK2982772 120 mg TID/240 mg TID/360 mg BID | Part A:GSK2982772 120 mg TID/240 mg TID/Placebo | Part A:GSK2982772 120 mg TID/Placebo/GSK2982772 360 mg BID | Part A:Placebo/GSK2982772 240 mg TID/360 mg BID | Part B:Placebo | Part B:GSK2982772 120 mg TID | Part B:GSK2982772 240 mg TID | Part B:GSK2982772 360 mg BID
Started | 3 (2 participants were added to GSK2982772 120 mg TID/240 mg TID/360 mg BID arm after Washout Period.) | 3 | 3 | 3 | 0 | 0 | 0 | 0
Completed | 3 | 3 | 3 | 3 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B (14 Days)
Arm/Group | Part A:GSK2982772 120 mg TID/240 mg TID/360 mg BID | Part A:GSK2982772 120 mg TID/240 mg TID/Placebo | Part A:GSK2982772 120 mg TID/Placebo/GSK2982772 360 mg BID | Part A:Placebo/GSK2982772 240 mg TID/360 mg BID | Part B:Placebo | Part B:GSK2982772 120 mg TID | Part B:GSK2982772 240 mg TID | Part B:GSK2982772 360 mg BID
Started | 0 | 0 | 0 | 0 | 14 | 20 | 13 | 0
Completed | 0 | 0 | 0 | 0 | 11 | 10 | 8 | 0
Not Completed | 0 | 0 | 0 | 0 | 3 | 10 | 5 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 2 | 4 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 2 | 8 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Participants were not enrolled into the GSK2982772 360 mg BID of Part B as one participant in the 360 mg BID dose level in Part A exceeded the maximum concentration (Cmax) stopping criteria.
Groups:
- Part A:GSK2982772 120 mg TID/240 mg TID/360 mg BID: Participants received oral capsule of 120 mg GSK2982772 three times a day in treatment period 1 followed by 240 mg TID in treatment period 2 followed by 360 mg BID in treatment period 3. The treatment periods were separated by a washout period of at least 7 days.
- Part B:GSK2982772 360 mg TID: Participants received GSK2982772 oral capsule at a dose of 360 mg TID for 14 days.
- Total: Total of all reporting groups
Arm/Group | Part A:GSK2982772 120 mg TID/240 mg TID/360 mg BID | Part A:GSK2982772 120 mg TID/240 mg TID/Placebo | Part A:GSK2982772 120 mg TID/Placebo/GSK2982772 360 mg BID | Part A:Placebo/GSK2982772 240 mg TID/360 mg BID | Part B:Placebo | Part B:GSK2982772 120 mg TID | Part B:GSK2982772 240 mg TID | Part B:GSK2982772 360 mg TID | Total
Number analyzed (Participants) | 5 | 4 | 3 | 3 | 14 | 20 | 13 | 0 | 62
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.2 (9.04) | 42.5 (9.95) | 59.0 (3.61) | 49.0 (10.00) | 39.1 (9.66) | 43.3 (10.87) | 38.6 (11.03) |  | 45.25 (9.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 5
  Male | 3 | 2 | 2 | 3 | 14 | 20 | 13 | 0 | 57
Race/Ethnicity, Customized [Number; unit: Participants]
  Black or African American | 0 | 1 | 1 | 0 | 0 | 1 | 3 |  | 6
  Asian - East Asian Heritage | 0 | 0 | 0 | 0 | 1 | 0 | 0 |  | 1
  Asian - Japanese Heritage | 0 | 0 | 0 | 0 | 1 | 0 | 0 |  | 1
  White - White/Caucasian/European Herit | 5 | 3 | 2 | 3 | 12 | 19 | 10 |  | 54

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Adverse Events (AEs) and Serious AEs (SAEs): Part A
Description: An AE is any untoward medical occurrence in a clinical study subjects, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect or any other situation according to medical or scientific judgment will be categorized as SAE.
Time Frame: Up to Day 14
Population: Safety population. Safety population consists of all randomized participants who take at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Part A:Placebo: Participants received matching oral placebo capsule to GSK2928772
- Part A:GSK2982772 120 mg TID: Participants received GSK2982772 oral capsule at a dose of 120 mg TID
- Part A:GSK2982772 240 mg TID: Participants received GSK2982772 oral capsule at a dose of 240 mg TID
- Part A:GSK2982772 360 mg BID: Participants received GSK2982772 oral capsule at a dose of 360 mg BID
Arm/Group | Part A:Placebo | Part A:GSK2982772 120 mg TID | Part A:GSK2982772 240 mg TID | Part A:GSK2982772 360 mg BID
Number analyzed (Participants) | 9 | 9 | 9 | 9
Participants
  AEs | 3 | 6 | 4 | 7
  SAEs | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With AEs and SAEs: Part B
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect or any other situation according to medical or scientific judgment were categorized as SAE.
Time Frame: Up to Day 28
Population: Safety population. GSK2982772 360 mg BID was not started in Part B as one participant in GSK2982772 360 mg BID of Part A exceeded the Cmax stopping criteria
Measure: Count of Participants; unit: Participants
Arm/Group | Part B:Placebo | Part B:GSK2982772 120 mg TID | Part B:GSK2982772 240 mg TID | Part B:GSK2982772 360 mg BID
Number analyzed (Participants) | 14 | 20 | 13 | 0
Participants
  AEs | 9 | 17 | 12 |
  SAEs | 1 | 0 | 0 |

3. Primary Outcome: Number of Participants With Worst Case Clinical Chemistry Parameters by Potential Clinical Importance Criteria: Part A
Description: Blood samples were collected from participants for the analysis of following clinical chemistry parameters: alanine amino transferase (ALT), albumin, alkaline phosphatase, aspartate amino transferase (AST), calcium, creatinine, glucose, potassium, sodium and total bilirubin. PCI ranges were >=2 times Upper Limit of Normal (ULN) units per liter (U/L) for ALT, <30 grams per liter (g/L) for albumin, >=2 times ULN U/L for alkaline phosphatase, >=2 times ULN U/L for AST, <2 or >2.75 millimoles per liter (mmol/L) for calcium, >44.2 micromoles per liter (µmol/L) for creatinine, <3 or >9 mmol/L for glucose, <3 or >5.5 mmol/L for potassium, <130 or >150 mmol/L for sodium and >=1.5 times ULN for total bilirubin. Participants were counted in the worst case category that their value changed to low, normal or high. If values were unchanged (example: High to High), or whose value became normal, were recorded in 'No Change' category.
Time Frame: Up to Week 9
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A:Placebo | Part A:GSK2982772 120 mg TID | Part A:GSK2982772 240 mg TID | Part A:GSK2982772 360 mg BID
Number analyzed (Participants) | 9 | 9 | 9 | 9
Participants
  ALT, Low | 0 | 0 | 0 | 0
  ALT, No change | 9 | 9 | 9 | 9
  ALT, High | 0 | 0 | 0 | 0
  Albumin, Low | 0 | 0 | 0 | 0
  Albumin, No change | 9 | 9 | 9 | 9
  Albumin, High | 0 | 0 | 0 | 0
  Alkaline phosphatase, Low | 0 | 0 | 0 | 0
  Alkaline phosphatase, No change | 9 | 9 | 9 | 9
  Alkaline phosphatase, High | 0 | 0 | 0 | 0
  AST, Low | 0 | 0 | 0 | 0
  AST, No change | 9 | 9 | 9 | 9
  AST, High | 0 | 0 | 0 | 0
  Calcium, Low | 0 | 0 | 0 | 0
  Calcium, No change | 9 | 9 | 9 | 9
  Calcium, High | 0 | 0 | 0 | 0
  Creatinine, Low | 0 | 0 | 0 | 0
  Creatinine, No change | 9 | 9 | 9 | 9
  Creatinine, High | 0 | 0 | 0 | 0
  Glucose, Low | 0 | 0 | 0 | 0
  Glucose, No change | 9 | 9 | 9 | 9
  Glucose, High | 0 | 0 | 0 | 0
  Potassium, Low | 0 | 0 | 0 | 0
  Potassium, No change | 9 | 9 | 9 | 9
  Potassium, High | 0 | 0 | 0 | 0
  Sodium, Low | 0 | 0 | 0 | 0
  Sodium, No change | 9 | 9 | 9 | 9
  Sodium, High | 0 | 0 | 0 | 0
  Total Bilirubin, Low | 0 | 0 | 0 | 0
  Total Bilirubin, No change | 9 | 9 | 9 | 9
  Total Bilirubin, High | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Worst Case Clinical Chemistry Parameters by Potential Clinical Importance Criteria: Part B
Description: Blood samples were collected from participants for the analysis of following clinical chemistry parameters: ALT, albumin, alkaline phosphatase, AST, calcium, creatinine, glucose, potassium, sodium and total bilirubin. PCI ranges were >=2 times ULN U/L for ALT, <30 g/L for albumin, >=2 times ULN U/L for alkaline phosphatase, >=2 times ULN U/L for AST, <2 or >2.75 mmol/L for calcium, >44.2 µmol/L for creatinine, <3 or >9 mmol/L for glucose, <3 or >5.5 mmol/L for potassium, <130 or >150 mmol/L for sodium and >=1.5 times ULN for total bilirubin. Participants were counted in the worst case category that their value changed to low, normal or high. If values were unchanged (example: High to High), or whose value became normal, were recorded in 'No Change' category.
Time Frame: Up to Week 4
Population: Safety population. GSK2982772 360 mg BID of Part B was not started as one participant in GSK2982772 360 mg BID of Part A exceeded the Cmax stopping criteria
Measure: Count of Participants; unit: Participants
Arm/Group | Part B:Placebo | Part B:GSK2982772 120 mg TID | Part B:GSK2982772 240 mg TID | Part B:GSK2982772 360 mg BID
Number analyzed (Participants) | 14 | 20 | 13 | 0
Participants
  ALT, Low | 0 | 0 | 0 |
  ALT, No change | 14 | 19 | 13 |
  ALT, High | 0 | 1 | 0 |
  Albumin, Low | 0 | 0 | 0 |
  Albumin, No change | 14 | 20 | 13 |
  Albumin, High | 0 | 0 | 0 |
  Alkaline phosphatase, Low | 0 | 0 | 0 |
  Alkaline phosphatase, No change | 14 | 20 | 13 |
  Alkaline phosphatase, High | 0 | 0 | 0 |
  AST, Low | 0 | 0 | 0 |
  AST, No change | 14 | 19 | 13 |
  AST, High | 0 | 1 | 0 |
  Calcium, Low | 0 | 0 | 0 |
  Calcium, No change | 14 | 20 | 13 |
  Calcium, High | 0 | 0 | 0 |
  Creatinine, Low | 0 | 0 | 0 |
  Creatinine, No change | 14 | 20 | 13 |
  Creatinine, High | 0 | 0 | 0 |
  Glucose, Low | 0 | 0 | 0 |
  Glucose, No change | 14 | 20 | 13 |
  Glucose, High | 0 | 0 | 0 |
  Potassium, Low | 0 | 0 | 0 |
  Potassium, No change | 14 | 20 | 12 |
  Potassium, High | 0 | 0 | 1 |
  Sodium, Low | 0 | 0 | 0 |
  Sodium, No change | 14 | 20 | 13 |
  Sodium, High | 0 | 0 | 0 |
  Total Bilirubin, Low | 0 | 0 | 0 |
  Total Bilirubin, No change | 14 | 20 | 13 |
  Total Bilirubin, High | 0 | 0 | 0 |

5. Primary Outcome: Number of Participants With Worst Case Hematology Parameters by Potential Clinical Importance Criteria: Part A
Description: Blood samples were collected from participants for analysis of following hematology parameters; hematocrit, hemoglobin, lymphocytes, platelet count, total neutrophils and white blood cell (WBC) counts. PCI ranges were >0.54 or < 0.075 proportion of red blood cells (RBC) in blood for hematocrit, <25 or >180 g/L for hemoglobin, 0.8 x10^9 cells/L for lymphocytes, <1.5 x10^9 cells/L for neutrophils, <100 or >550 x10^9 cells/L for platelets and <3 or 20> x 10^9 cells per liter WBC. Participants were counted in the worst case category that their value changed to low, normal or high. If values were unchanged (example: High to High), or whose value became normal, were recorded in 'No Change' category.
Time Frame: Up to Week 9
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A:Placebo | Part A:GSK2982772 120 mg TID | Part A:GSK2982772 240 mg TID | Part A:GSK2982772 360 mg BID
Number analyzed (Participants) | 9 | 9 | 9 | 9
Participants
  Hematocrit, Low | 0 | 0 | 0 | 0
  Hematocrit, No change | 9 | 9 | 9 | 9
  Hematocrit, High | 0 | 0 | 0 | 0
  Hemoglobin, Low | 0 | 0 | 0 | 0
  Hemoglobin, No change | 9 | 9 | 9 | 9
  Hemoglobin, High | 0 | 0 | 0 | 0
  Lymphocytes, Low | 0 | 0 | 0 | 0
  Lymphocytes, No change | 9 | 9 | 9 | 9
  Lymphocytes, High | 0 | 0 | 0 | 0
  Platelet count, Low | 0 | 0 | 0 | 0
  Platelet, No change | 9 | 9 | 9 | 9
  Platelet, High | 0 | 0 | 0 | 0
  Total Neutrophils, Low | 1 | 0 | 0 | 0
  Total Neutrophils, No change | 8 | 9 | 9 | 9
  Total Neutrophils, High | 0 | 0 | 0 | 0
  WBC count, Low | 0 | 0 | 0 | 0
  WBC, No change | 9 | 9 | 9 | 9
  WBC, High | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Participants With Worst Case Hematology Parameters by Potential Clinical Importance Criteria: Part B
Description: Blood samples were collected from participants for analysis of following hematology parameters; hematocrit, hemoglobin, lymphocytes, platelet count, total neutrophils and WBC counts. PCI ranges were >0.54 or < 0.075 proportion of RBC in blood for hematocrit, <25 or >180 g/L for hemoglobin, 0.8 x10^9 cells/L for lymphocytes, <1.5 x10^9 cells/L for neutrophils, <100 or >550 x10^9 cells/L for platelets and <3 or 20> x 10^9 cells per liter WBC. Participants were counted in the worst case category that their value changed to low, normal or high. If values were unchanged (example: High to High), or whose value became normal, were recorded in 'No Change' category.
Time Frame: Up to Week 4
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Part B:Placebo | Part B:GSK2982772 120 mg TID | Part B:GSK2982772 240 mg TID | Part B:GSK2982772 360 mg BID
Number analyzed (Participants) | 14 | 20 | 13 | 0
Participants
  Hematocrit, Low | 0 | 0 | 0 |
  Hematocrit, No change | 14 | 20 | 13 |
  Hematocrit, High | 0 | 0 | 0 |
  Hemoglobin, Low | 0 | 0 | 0 |
  Hemoglobin, No change | 14 | 20 | 13 |
  Hemoglobin, High | 0 | 0 | 0 |
  Lymphocytes, Low | 0 | 0 | 1 |
  Lymphocytes, No change | 14 | 20 | 12 |
  Lymphocytes, High | 0 | 0 | 0 |
  Platelet count, Low | 0 | 0 | 0 |
  Platelet, No change | 14 | 20 | 13 |
  Platelet, High | 0 | 0 | 0 |
  Total Neutrophils, Low | 0 | 1 | 3 |
  Total Neutrophils, No change | 14 | 19 | 10 |
  Total Neutrophils, High | 0 | 0 | 0 |
  WBC count, Low | 0 | 0 | 0 |
  WBC, No change | 14 | 20 | 13 |
  WBC, High | 0 | 0 | 0 |

7. Primary Outcome: Number of Participants With Worst Case Urinalysis Results: Part A
Description: Urine samples were collected from participants for analysis of following parameters: cellular casts, granular casts, hyaline casts, RBC and WBC and were counted as cells per high-power field (cells/HPF). The number of participants with cells in urine has been presented.
Time Frame: Up to Week 9
Population: Safety population. Only those participants with available data at specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A:Placebo | Part A:GSK2982772 120 mg TID | Part A:GSK2982772 240 mg TID | Part A:GSK2982772 360 mg BID
Number analyzed (Participants) | 3 | 1 | 1 | 1
Participants
  Cellular casts, No change | 3 | 1 | 1 | 1
  Cellular casts, Any increase | 0 | 0 | 0 | 0
  Cellular casts, Increase to 1-9/HPF | 0 | 0 | 0 | 0
  Cellular casts, Increase to 10-50/HPF | 0 | 0 | 0 | 0
  Granular casts, No change | 3 | 1 | 1 | 1
  Granular casts, Any increase | 0 | 0 | 0 | 0
  Granular casts, Increase 1-9/HPF | 0 | 0 | 0 | 0
  Granular casts, Increase 10-50/HPF | 0 | 0 | 0 | 0
  Hyaline casts, No change | 3 | 1 | 1 | 1
  Hyaline casts, Any increase | 0 | 0 | 0 | 0
  Hyaline casts, Increase 1-9/HPF | 0 | 0 | 0 | 0
  Hyaline casts, Increase 10-50/HPF | 0 | 0 | 0 | 0
  RBC, No change | 3 | 0 | 1 | 0
  RBC, Any increase | 0 | 1 | 0 | 1
  RBC, Increase 1-9/HPF | 0 | 1 | 0 | 1
  RBC, Increase 10-50/HPF | 0 | 0 | 0 | 0
  WBC, No change | 3 | 1 | 1 | 0
  WBC, Any increase | 0 | 0 | 0 | 1
  WBC, Increase 1-9/HPF | 0 | 0 | 0 | 1
  WBC, Increase 10-50/HPF | 0 | 0 | 0 | 0

8. Primary Outcome: Number of Participants With Worst Case Urinalysis Results: Part B
Description: as for outcome 7
Time Frame: Up to Week 4
Population: Safety population. GSK2982772 360 mg BID of Part B was not started as one participant in GSK2982772 360 mg BID of Part A exceeded the Cmax stopping criteria. Only those participants with data available at specified timepoints were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B:Placebo | Part B:GSK2982772 120 mg TID | Part B:GSK2982772 240 mg TID | Part B:GSK2982772 360 mg BID
Number analyzed (Participants) | 0 | 7 | 2 | 0
Participants
  Cellular casts, No change |  | 7 | 2 |
  Cellular casts, Any increase |  | 0 | 0 |
  Cellular casts, Increase to 1-9/HPF |  | 0 | 0 |
  Cellular casts, Increase to 10-50/HPF |  | 0 | 0 |
  Granular casts, No change |  | 7 | 2 |
  Granular casts, Any increase |  | 0 | 0 |
  Granular casts, Increase 1-9/HPF |  | 0 | 0 |
  Granular casts, Increase 10-50/HPF |  | 0 | 0 |
  Hyaline casts, No change |  | 7 | 2 |
  Hyaline casts, Any increase |  | 0 | 0 |
  Hyaline casts, Increase 1-9/HPF |  | 0 | 0 |
  Hyaline casts, Increase 10-50/HPF |  | 0 | 0 |
  RBC, No change |  | 5 | 1 |
  RBC, Any increase |  | 2 | 1 |
  RBC, Increase 1-9/HPF |  | 2 | 1 |
  RBC, Increase 10-50/HPF |  | 0 | 0 |
  WBC, No change |  | 5 | 2 |
  WBC, Any increase |  | 2 | 0 |
  WBC, Increase 1-9/HPF |  | 2 | 0 |
  WBC, Increase 10-50/HPF |  | 0 | 0 |

9. Primary Outcome: Number of Participants With Abnormal Vital Signs: Part A
Description: Vital signs were measured in a supine position after 5 minutes rest. The PCI criteria for vital signs included: systolic blood pressure <85 and >160 millimeters of mercury [mmHg]), diastolic blood pressure <45 mmHg and >100 mmHg, heart rate <40 and >100 beats per minute, body temperature <=35.5 and >=37.8 degrees Celsius and respiration rate <=8 and >=20 breaths per minute. Data of participants with potential clinical importance has been reported.
Time Frame: Up to Week 9
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A:Placebo | Part A:GSK2982772 120 mg TID | Part A:GSK2982772 240 mg TID | Part A:GSK2982772 360 mg BID
Number analyzed (Participants) | 9 | 9 | 9 | 9
Participants | 6 | 8 | 7 | 8

10. Primary Outcome: Number of Participants With Abnormal Vital Signs: Part B
Description: Vital signs were measured in a supine position after 5 minutes rest. The PCI criteria for vital signs included: systolic blood pressure <85 and >160 mmHg, diastolic blood pressure <45 mmHg and >100 mmHg, heart rate <40 and >100 beats per minute, body temperature <=35.5 and >=37.8 degrees Celsius and respiration rate <=8 and >=20 breaths per minute. Data of participants with potential clinical importance has been reported.
Time Frame: Up to Week 4
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Part B:Placebo | Part B:GSK2982772 120 mg TID | Part B:GSK2982772 240 mg TID | Part B:GSK2982772 360 mg BID
Number analyzed (Participants) | 14 | 20 | 13 | 0
Participants | 11 | 20 | 12 |

11. Primary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Findings: Part A
Description: 12-lead ECG's were obtained in the supine position after 5 minutes of rest using an ECG machine that automatically calculated the heart rate and measured PR, QRS, QT and QT duration corrected for heart rate by Fridericia's formula (QTcF) intervals. Clinically significant and not clinically significant abnormal ECG findings have been presented. Clinically significant abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
Time Frame: Up to Day 4
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A:Placebo | Part A:GSK2982772 120 mg TID | Part A:GSK2982772 240 mg TID | Part A:GSK2982772 360 mg BID
Number analyzed (Participants) | 9 | 9 | 9 | 9
Participants
  Abnormal, not clinically significant | 1 | 0 | 2 | 4
  Abnormal, clinically significant | 0 | 0 | 0 | 0

12. Primary Outcome: Number of Participants With Abnormal ECG Findings: Part B
Description: as for outcome 11
Time Frame: Up to Week 4
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Part B:Placebo | Part B:GSK2982772 120 mg TID | Part B:GSK2982772 240 mg TID | Part B:GSK2982772 360 mg BID
Number analyzed (Participants) | 14 | 20 | 13 | 0
Participants
  Abnormal, not clinically significant | 3 | 4 | 3 |
  Abnormal, clinically significant | 0 | 0 | 0 |

13. Secondary Outcome: Area Under the Concentration-time Curve (AUC) From Time Zero to 24 Hours (AUC[0-24]) Following TID Dosing of GSK2982772: Part A
Description: Blood samples were collected at indicated timepoints for pharmacokinetic analysis of GSK2982772. Pharmacokinetic parameters were calculated by standard non-compartmental analysis.
Time Frame: Pre-dose, 20, 40minutes, 1 hour, 1hr 30min, 2, 3, 5, 7hour, 7hr 20min,and 7hr 40 min, 8hr, 8hr 30min, 9hr, 10hr, 12hr, 14hr, 14hr 20min, 14hr 40 min, 15hr, 15hr 30min, 16hr, 17hr, 19hr, 22hr, 24hours post dose on Day1
Population: Pharmacokinetic population. Pharmacokinetic population consists of participants in the safety population for whom a pharmacokinetic sample were obtained and analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per millilter
Arm/Group | Part A:GSK2982772 120 mg TID | Part A:GSK2982772 240 mg TID
Number analyzed (Participants) | 9 | 9
Hours*microgram per millilter | 21.22 (41.37) | 46.13 (37.38)

14. Secondary Outcome: AUC(0-24) Following BID Dosing of GSK2982772: Part A
Description: as for outcome 13
Time Frame: Pre-dose, 20min, 40min, 1hr, 1hr 30min, 2hr, 3hr, 4hr, 6hr, 8hr, 10hr, 12hr, 12hr 20min, 12hr 40min, 13hr, 13hr 30min, 14hr, 15hr, 16hr, 19hr, 22hr, 24hr post dose on Day 1.
Population: Pharmacokinetic population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per millilter
Arm/Group | Part A:GSK2982772 360 mg BID
Number analyzed (Participants) | 9
Hours*microgram per millilter | 54.02 (36.02)

15. Secondary Outcome: AUC[0-24] Following TID Dosing of GSK2982772: Part B
Description: as for outcome 13
Time Frame: Pre-dose, 20, 40minutes, 1 hour, 1hr 30min, 2, 3, 5, 7hour, 7hr 20min,and 7hr 40 min, 8hr, 8hr 30min, 9hr, 10hr, 12hr, 14hr, 14hr 20min, 14hr 40 min, 15hr, 15hr 30min, 16hr, 17hr, 19hr, 22hr, 24hours post dose on Day14
Population: Pharmacokinetic population. Only those participants with data available at the specified timepoints were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per millilter
Arm/Group | Part B:GSK2982772 120 mg TID | Part B:GSK2982772 240 mg TID
Number analyzed (Participants) | 10 | 8
Hours*microgram per millilter | 25.67 (28.81) | 52.00 (45.26)

16. Secondary Outcome: AUC (0-7) Following TID Dosing of GSK2982772 : Part A
Description: as for outcome 13
Time Frame: Pre-dose, 20 and 40 minutes, 1 and 1 hour 30 minutes, 2, 3, 5, 7 hours on Day 1
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per millilter
Arm/Group | Part A:GSK2982772 120 mg TID | Part A:GSK2982772 240 mg TID
Number analyzed (Participants) | 9 | 9
Hours*microgram per millilter | 6.053 (33.87) | 11.686 (33.50)

17. Secondary Outcome: AUC (7-14) Following TID Dosing of GSK2982772 : Part A
Description: as for outcome 13
Time Frame: 7 hours, 7 hours 20 and 40 minutes, 8 hours, 8 hours 30 minutes, 9, 10, 12, 14 hours on Day 1
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per millilter
Arm/Group | Part A:GSK2982772 120 mg TID | Part A:GSK2982772 240 mg TID
Number analyzed (Participants) | 9 | 9
Hours*microgram per millilter | 7.829 (44.25) | 17.823 (42.11)

18. Secondary Outcome: AUC (14-24) Following TID Dosing of GSK2982772 : Part A
Description: as for outcome 13
Time Frame: 14 hours, 14 hours 20 and 40 minutes, 15 hours ,15 hours 30 minutes, 16, 19, 22 and 24 hours on Day 1
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per millilter
Arm/Group | Part A:GSK2982772 120 mg TID | Part A:GSK2982772 240 mg TID
Number analyzed (Participants) | 9 | 9
Hours*microgram per millilter | 7.213 (48.85) | 16.300 (39.72)

19. Secondary Outcome: AUC (0-12) Following BID Dosing of GSK2982772 in Part A
Description: as for outcome 13
Time Frame: Pre-dose, 20 and 40 minutes, 1 and 1 hour 30 minutes, 2, 3, 4, 6, 8, 10 hours,12 hours on Day 1
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per millilter
Arm/Group | Part A:GSK2982772 360 mg BID
Number analyzed (Participants) | 9
Hours*microgram per millilter | 21.80 (24.41)

20. Secondary Outcome: AUC (12-24) Following BID Dosing of GSK2982772 in Part A
Description: as for outcome 13
Time Frame: 12 hours, 12 hours 20 and 40 minutes, 13 and 13 hours 30 minutes, 14, 15, 16, 19, 22 and 24 hours on Day 1
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per millilter
Arm/Group | Part A:GSK2982772 360 mg BID
Number analyzed (Participants) | 9
Hours*microgram per millilter | 31.69 (48.02)

21. Secondary Outcome: AUC(0-7) Following TID Dosing of GSK2982772 in Part B
Description: Blood samples were collected at indicated time-points for pharmacokinetic analysis of GSK2982772. Pharmacokinetic parameters were calculated by standard non-compartmental analysis.
Time Frame: Pre-dose, 20 and 40 minutes, 1 and 1 hour 30 minutes, 2, 3, 5, 7 hours on Days 1 and 14
Population: Pharmacokinetic population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*microgram per millilter
Arm/Group | Part B:GSK2982772 120 mg TID | Part B:GSK2982772 240 mg TID
Number analyzed (Participants) | 20 | 13
Hour*microgram per millilter
  AUC (0-7), Day 1, n=20, 13 | 6.550 (37.67) | 11.895 (33.98)
  AUC (0-7), Day 14, n=10, 9: number analyzed (Participants) | 10 | 9
  AUC (0-7), Day 14, n=10, 9 | 7.485 (25.53) | 14.835 (45.30)

22. Secondary Outcome: AUC (7-14) Following TID Dosing of GSK2982772 in Part B
Description: as for outcome 21
Time Frame: 7 and 7 hours 20 and 40 minutes, 8 and 8 hours 30 minutes, 9, 10, 12, 14 hours on Day 14
Population: Pharmacokinetic population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per millilter
Arm/Group | Part B:GSK2982772 120 mg TID | Part B:GSK2982772 240 mg TID
Number analyzed (Participants) | 10 | 8
Hours*microgram per millilter | 9.095 (30.57) | 17.372 (34.96)

23. Secondary Outcome: AUC (14-24) Following TID Dosing of GSK2982772 in Part B
Description: as for outcome 21
Time Frame: 14 hours, 14 hours 20 minutes, 14 hours 40 minutes, 15 hours, 15 hours 30 minutes, 16, 17, 19, 22 and 24 hours on Day 14
Population: Pharmacokinetic population. Only those participants with data available at the specified data points were analyzed
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per millilter
Arm/Group | Part B:GSK2982772 120 mg TID | Part B:GSK2982772 240 mg TID
Number analyzed (Participants) | 10 | 8
Hours*microgram per millilter | 8.988 (33.57) | 19.816 (55.60)

24. Secondary Outcome: Maximum Observed Plasma Drug Concentration Cmax (0-7) Following TID Dosing of GSK2982772 in Part A
Description: as for outcome 21
Time Frame: Pre-dose, 20 and 40 minutes, 1 and 1 hour 30 minutes, 2, 3, 5, and 7 hours post dose on Day 1
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Part A:GSK2982772 120 mg TID | Part A:GSK2982772 240 mg TID
Number analyzed (Participants) | 9 | 9
Microgram per milliliter | 1.7672 (41.78) | 3.3125 (25.88)

25. Secondary Outcome: Cmax (7-14) Following TID Dosing of GSK2982772 in Part A
Description: as for outcome 21
Time Frame: 7 hours, 7 hours 20 and 40 minutes, 8 and 8 hours 30 minutes, 9, 10, 12, 14 hours post dose on Day 1
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Part A:GSK2982772 120 mg TID | Part A:GSK2982772 240 mg TID
Number analyzed (Participants) | 9 | 9
Microgram per milliliter | 2.148 (36.24) | 5.007 (33.09)

26. Secondary Outcome: Cmax (14-24) Following TID Dosing of GSK2982772 in Part A
Description: as for outcome 21
Time Frame: 14 hours, 14 hours 20 and 40 minutes, 15 and 15 hours 30 minutes, 16, 19, 22 and 24 hours post dose on Day 1
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Part A:GSK2982772 120 mg TID | Part A:GSK2982772 240 mg TID
Number analyzed (Participants) | 9 | 9
Microgram per milliliter | 1.4156 (47.03) | 3.4812 (28.46)

27. Secondary Outcome: Cmax (0-12) Following BID Dosing of GSK2982772 in Part A
Description: as for outcome 21
Time Frame: Pre-dose, 20 and 40 minutes, 1 and 1 hour 30 minutes, 2, 3, 4, 6, 8, 10 hours and 12 hours post dose on Day 1
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Part A:GSK2982772 360 mg BID
Number analyzed (Participants) | 9
Microgram per milliliter | 4.967 (30.75)

28. Secondary Outcome: Cmax (12-24) Following BID Dosing of GSK2982772 in Part A
Description: as for outcome 21
Time Frame: 12 hours, 12 hours 20 and 40 minutes, 13 and 13 hours 30 minutes, 14, 15, 16, 19, 22 and 24 hours post dose on Day 1
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Part A:GSK2982772 360 mg BID
Number analyzed (Participants) | 9
Microgram per milliliter | 6.965 (61.70)

29. Secondary Outcome: Cmax (0-7) Following TID Dosing of GSK2982772 in Part B
Description: as for outcome 21
Time Frame: Pre-dose, 20 and 40 minutes, 1 and 1 hour 30 minutes, 2, 3, 5, 7 hours post dose on Days 1 and 14
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Part B:GSK2982772 120 mg TID | Part B:GSK2982772 240 mg TID
Number analyzed (Participants) | 20 | 13
Microgram per milliliter
  Cmax (0-7), Day 1, n=20, 13 | 2.0883 (37.87) | 3.2333 (37.04)
  Cmax (0-7), Day 14, n=10, 9: number analyzed (Participants) | 10 | 9
  Cmax (0-7), Day 14, n=10, 9 | 2.2239 (30.03) | 4.3784 (45.62)

30. Secondary Outcome: Cmax (7-14) Following TID Dosing of GSK2982772 in Part B
Description: as for outcome 21
Time Frame: 7hours, 7 hours 20 and 40 minutes, 8 hours, 8 hours 30 minutes, 9, 10, 12, 14 hours on Day 14
Population: Pharmacokinetic population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Part B:GSK2982772 120 mg TID | Part B:GSK2982772 240 mg TID
Number analyzed (Participants) | 10 | 8
Microgram per milliliter | 2.505 (26.70) | 5.435 (32.59)

31. Secondary Outcome: Cmax (14-24) Following TID Dosing of GSK2982772 in Part B
Description: as for outcome 21
Time Frame: 14 hours, 14 hours 20 and 40 minutes, 15 hours, 15 hours 30 minutes, 16, 17, 19, 22 and 24 hours post dose on Day 14
Population: Pharmacokinetic population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per millilter
Arm/Group | Part B:GSK2982772 120 mg TID | Part B:GSK2982772 240 mg TID
Number analyzed (Participants) | 10 | 8
Microgram per millilter | 1.9205 (30.82) | 4.1607 (38.79)

32. Secondary Outcome: Time to Cmax (Tmax) (0-7) Following TID Dosing of GSK2982772 in Part A
Description: as for outcome 21
Time Frame: Pre-dose, 20 and 40 minutes, 1 and 1 hour 30 minutes, 2, 3, 5, and 7 hours post dose on Day 1
Population: Pharmacokinetic population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A:GSK2982772 120 mg TID | Part A:GSK2982772 240 mg TID
Number analyzed (Participants) | 9 | 9
Hours | 3.008 [2.00 to 5.02] | 2.043 [1.50 to 3.01]

33. Secondary Outcome: Tmax (7-14) Following TID Dosing of GSK2982772 in Part A
Description: as for outcome 21
Time Frame: 7hours, 7 hours 20 and 40 minutes, 8 hours, 8 hours 30 minutes, 9, 10, 12, 14 hours post dose on Day 1
Population: Pharmacokinetic population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A:GSK2982772 120 mg TID | Part A:GSK2982772 240 mg TID
Number analyzed (Participants) | 9 | 9
Hours | 10.000 [8.00 to 12.00] | 9.000 [8.50 to 10.02]

34. Secondary Outcome: Tmax (14-24) Following TID Dosing of GSK2982772 in Part A
Description: as for outcome 21
Time Frame: 14 hours, 14 hours 20 and 40 minutes, 15 hours, 15 hours 30 minutes, 16, 17, 19, 22 and 24 hours post dose on Day 1
Population: Pharmacokinetic population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A:GSK2982772 120 mg TID | Part A:GSK2982772 240 mg TID
Number analyzed (Participants) | 9 | 9
Hours | 19.00 [16.0 to 22.0] | 17.02 [16.0 to 24.0]

35. Secondary Outcome: Tmax (0-12) Following BID Dosing of GSK2982772 in Part A
Description: as for outcome 21
Time Frame: Pre-dose, 20 and 40 minutes, 1hour, 1 hour 30 minutes, 2, 3, 4, 6, 8, 10 hours and 12 hours post dose on Day 1
Population: Pharmacokinetic population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A:GSK2982772 360 mg BID
Number analyzed (Participants) | 9
Hours | 3.000 [1.50 to 4.02]

36. Secondary Outcome: Tmax (12-24) Following BID Dosing of GSK2982772 in Part A
Description: Blood samples were collected at indicated time-points for pharmacokinetic analysis of GSK2982772.Pharmacokinetic parameters were calculated by standard non-compartmental analysis.
Time Frame: 12 hours, 12 hours 20 and 40 minutes, 13 hours, 13 hours 30 minutes, 14, 15, 16, 19, 22 and 24 hours post dose on Day 1
Population: Pharmacokinetic population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A:GSK2982772 360 mg BID
Number analyzed (Participants) | 9
Hours | 14.01 [13.5 to 15.0]

37. Secondary Outcome: Tmax (0-7) Following TID Dosing of GSK2982772 Part B
Description: as for outcome 21
Time Frame: Pre-dose, 20 and 40 minutes, 1 hour, 1 hour 30 minutes, 2, 3, 5, 7 hours post dose on Days 1 and 14
Population: as for outcome 21
Measure: Median (Full Range); unit: Hours
Arm/Group | Part B:GSK2982772 120 mg TID | Part B:GSK2982772 240 mg TID
Number analyzed (Participants) | 20 | 13
Hours
  Tmax (0-7), Day 1, n=20, 13 | 2.000 [1.00 to 3.01] | 3.000 [1.00 to 3.01]
  Tmax (0-7), Day 14, n=10, 9: number analyzed (Participants) | 10 | 9
  Tmax (0-7), Day 14, n=10, 9 | 1.750 [1.00 to 3.03] | 2.003 [1.00 to 3.00]

38. Secondary Outcome: Tmax (7-14) Following TID Dosing of GSK2982772 in Part B
Description: as for outcome 21
Time Frame: 7hours and 7 hours 20 and 40 minutes, 8hours, 8 hours 30 minutes, 9, 10, 12, 14 hours post dose on Day 14
Population: Pharmacokinetic population. Only those participants with data available at the specified data points were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part B:GSK2982772 120 mg TID | Part B:GSK2982772 240 mg TID
Number analyzed (Participants) | 10 | 8
Hours | 9.001 [8.50 to 10.00] | 10.008 [8.50 to 12.00]

39. Secondary Outcome: Tmax (14-24) Following TID Dosing of GSK2982772 in Part B
Description: as for outcome 21
Time Frame: 14hours, 14 hours 20 and 40 minutes, 15 hours and 15 hours 30 minutes, 16, 17, 19, 22 and 24 hours post dose on Day 14
Population: Pharmacokinetic population. Only those participants with data available at the specified data points were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part B:GSK2982772 120 mg TID | Part B:GSK2982772 240 mg TID
Number analyzed (Participants) | 10 | 8
Hours | 17.02 [15.0 to 19.0] | 18.92 [16.0 to 19.0]

40. Secondary Outcome: Observed Trough Plasma Drug Concentration at 7 Hour (C7),Following TID Dosing of GSK2982772 in Part A
Description: as for outcome 21
Time Frame: 7 hours post-dose on Day 1
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Part A:GSK2982772 120 mg TID | Part A:GSK2982772 240 mg TID
Number analyzed (Participants) | 9 | 9
Microgram per milliliter | 0.3614 (84.67) | 0.7723 (89.30)

41. Secondary Outcome: Observed Trough Plasma Drug Concentration at 14 Hours (C14) Following TID Dosing of GSK2982772 in Part A
Description: as for outcome 21
Time Frame: 14 hours post-dose on Day 1
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Part A:GSK2982772 120 mg TID | Part A:GSK2982772 240 mg TID
Number analyzed (Participants) | 9 | 9
Microgram per milliliter | 0.4318 (86.28) | 0.7487 (76.95)

42. Secondary Outcome: C24 Following TID Dosing of GSK2982772 in Part A
Description: as for outcome 21
Time Frame: 24 hours post-dose on Day 1
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Part A:GSK2982772 120 mg TID | Part A:GSK2982772 240 mg TID
Number analyzed (Participants) | 9 | 9
Microgram per milliliter | 0.34518 (82.34) | 0.59880 (158.88)

43. Secondary Outcome: C12 Following BID Dosing of GSK2982772 in Part A
Description: Blood samples were collected at indicated time-points for pharmacokinetic analysis of GSK2982772.Pharmacokinetic parameters were calculated by standard non-compartmental analysis.
  Pharmacokinetic parameters were calculated by standard non-compartmental analysis.
Time Frame: 12 hours post-dose on Day 1
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per millilter
Arm/Group | Part A:GSK2982772 360 mg BID
Number analyzed (Participants) | 9
Microgram per millilter | 0.3490 (98.83)

44. Secondary Outcome: C24 Following BID Dosing of GSK2982772 in Part A
Description: as for outcome 36
Time Frame: 24 hours post-dose on Day 1
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per millililter
Arm/Group | Part A:GSK2982772 360 mg BID
Number analyzed (Participants) | 9
Microgram per millililter | 0.36965 (101.70)

45. Secondary Outcome: C0 Following TID Dosing of GSK2982772 in Part B
Description: as for outcome 36
Time Frame: Pre-dose on Day 14
Population: Pharmacokinetic population. Only those participants with data available at the specified data points were analyzed
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Part B:GSK2982772 120 mg TID | Part B:GSK2982772 240 mg TID
Number analyzed (Participants) | 10 | 8
Microgram per milliliter | 0.29926 (56.63) | 0.57528 (136.34)

46. Secondary Outcome: C7 Following TID Dosing of GSK2982772 in Part B
Description: as for outcome 36
Time Frame: 7 hours post-dose on Days 1 and 14
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Part B:GSK2982772 120 mg TID | Part B:GSK2982772 240 mg TID
Number analyzed (Participants) | 20 | 13
Microgram per milliliter
  C7, Day 1, n=20, 13 | 0.3345 (50.78) | 0.6105 (57.01)
  C7, Day 14, n=10, 9: number analyzed (Participants) | 10 | 9
  C7, Day 14, n=10, 9 | 0.3718 (43.85) | 0.6885 (75.98)

47. Secondary Outcome: C14 Following TID Dosing of GSK2982772 in Part B
Description: as for outcome 36
Time Frame: 14 hours post-dose on Day 14
Population: Pharmacokinetic population. Only those participants with data available at the specified data points were analyzed
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Part B:GSK2982772 120 mg TID | Part B:GSK2982772 240 mg TID
Number analyzed (Participants) | 10 | 9
Microgram per milliliter | 0.3830 (53.04) | 0.6912 (106.01)

48. Secondary Outcome: C24 Following TID Dosing of GSK2982772 in Part B
Description: as for outcome 36
Time Frame: 24 hours post-dose on Day 14
Population: Pharmacokinetic population. Only those participants with data available at the specified data points were analyzed
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Part B:GSK2982772 120 mg TID | Part B:GSK2982772 240 mg TID
Number analyzed (Participants) | 10 | 9
Microgram per milliliter | 0.22712 (60.78) | 0.33342 (180.82)

49. Secondary Outcome: AUC([0-7] Following TID Dosing of GSK2982772 in Fed State of Part B
Description: as for outcome 36
Time Frame: Pre-dose, 20 and 40 minutes, 1 and 1 hour 30 minutes, 2, 3, 5, 7 hours on Days 9 and 11
Population: Pharmacokinetic population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | Part B:GSK2982772 120 mg TID | Part B:GSK2982772 240 mg TID
Number analyzed (Participants) | 14 | 9
Hours*micrograms per milliliter
  AUC (0-7) following normal breakfast, Day 9 | 7.743 (31.46) | 14.691 (37.63)
  AUC (0-7) following high fat breakfast, Day 11 | 6.874 (24.64) | 15.987 (42.86)

50. Secondary Outcome: Cmax (0-7) Following TID Dosing of GSK2982772 in Fed State of Part B
Description: as for outcome 36
Time Frame: Pre-dose, 20 and 40 minutes, 1 and 1 hour 30 minutes, 2, 3, 5, 7 hours on Days 9 and 11
Population: Pharmacokinetic population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Part B:GSK2982772 120 mg TID | Part B:GSK2982772 240 mg TID
Number analyzed (Participants) | 14 | 9
Microgram per milliliter
  Cmax(0-7), following Normal Breakfast, Day 9 | 2.0918 (21.74) | 3.9440 (33.82)
  Cmax(0-7), following High Fat Breakfast, Day 11 | 1.8098 (29.77) | 4.1171 (58.36)

51. Secondary Outcome: Tmax (0-7) Following TID Dosing of GSK2982772 in Fed State of Part B
Description: as for outcome 36
Time Frame: Pre-dose, 20 and 40 minutes, 1 and 1 hour 30 minutes, 2, 3, 5, 7 hours on Days 9 and 11
Population: Pharmacokinetic population. Only those participants with data available at the specified data points were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part B:GSK2982772 120 mg TID | Part B:GSK2982772 240 mg TID
Number analyzed (Participants) | 14 | 9
Hours
  Tmax(0-7), Day 9 | 3.000 [1.04 to 5.00] | 3.000 [2.00 to 5.03]
  Tmax (0-7), Day 11 | 4.000 [1.50 to 5.00] | 3.000 [2.00 to 5.00]

52. Secondary Outcome: Ratio of Plasma 4 Beta-hydroxycholesterol to Cholesterol: Part B
Description: Blood samples were collected into EDTA tubes and processed to plasma for 4 beta-hydroxycholesterol and cholesterol. Ratio of 4 beta-hydroxycholesterol to cholesterol is presented
Time Frame: Pre-dose on Day 1 and 24 hours post first dose on Day 14
Population: Pharmacokinetic population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part B:Placebo | Part B:GSK2982772 120 mg TID | Part B:GSK2982772 240 mg TID
Number analyzed (Participants) | 1 | 20 | 13
Ratio
  Day 1, Pre-dose; n=0, 19, 12: number analyzed (Participants) | 0 | 19 | 12
  Day 1, Pre-dose; n=0, 19, 12 |  | 0.000019 (0.0000064) | 0.000023 (0.0000099)
  Day 14, 24 hour; n=1, 10, 9: number analyzed (Participants) | 1 | 10 | 9
  Day 14, 24 hour; n=1, 10, 9 | 0.000016 (NA) — Not applicable (NA) indicates that standard deviation could not be calculated for a single participant. | 0.000021 (0.0000089) | 0.000024 (0.0000065)

ADVERSE EVENTS:
Time Frame: On-treatment SAEs and non serious AEs were collected from the start of study treatment up to Day 14 for Part A and up to Day 28 for Part B.
Description: Safety population consists of all randomized participants who take at least 1 dose of study treatment.
Groups:
- Part A: Placebo: Participants received matching oral placebo capsule to GSK2928772
- Part A: GSK2982772 240 mg TID: Participants received GSK2982772 oral capsule at a dose of 240 mg TID
- Part A: GSK2982772 360 mg BID: Participants received GSK2982772 oral capsule at a dose of 360 mg BID
- Part B: GSK2982772 120 mg TID: Participants received GSK2982772 oral capsule at a dose of 120 mg TID for 14 days
- Part B: GSK2982772 240 mg TID: Participants received GSK2982772 oral capsule at a dose of 240 mg TID for 14 days
- Part B: GSK2982772 360 mg BID: Participants were planned to receive GSK2982772 oral capsule at a dose of 360 mg TID for 14 days
Arm/Group | Part A: Placebo | Part A:GSK2982772 120 mg TID | Part A: GSK2982772 240 mg TID | Part A: GSK2982772 360 mg BID | Part B:Placebo | Part B: GSK2982772 120 mg TID | Part B: GSK2982772 240 mg TID | Part B: GSK2982772 360 mg BID
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/9 | 0/14 | 0/20 | 0/13 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/9 | 1/14 | 0/20 | 0/13 | 0/0
Other Adverse Events (participants affected / at risk) | 3/9 | 6/9 | 4/9 | 7/9 | 9/14 | 17/20 | 12/13 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Placebo (N=9) | Part A:GSK2982772 120 mg TID (N=9) | Part A: GSK2982772 240 mg TID (N=9) | Part A: GSK2982772 360 mg BID (N=9) | Part B:Placebo (N=14) | Part B: GSK2982772 120 mg TID (N=20) | Part B: GSK2982772 240 mg TID (N=13) | Part B: GSK2982772 360 mg BID (N=0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Placebo (N=9) | Part A:GSK2982772 120 mg TID (N=9) | Part A: GSK2982772 240 mg TID (N=9) | Part A: GSK2982772 360 mg BID (N=9) | Part B:Placebo (N=14) | Part B: GSK2982772 120 mg TID (N=20) | Part B: GSK2982772 240 mg TID (N=13) | Part B: GSK2982772 360 mg BID (N=0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 3 (3) | 3 (3) | 3 (4) | 4 (4) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Faeces soft (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medical device site dermatitis (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thirst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 4 (4) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Catheter site bruise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mood altered (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nightmare (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Polyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear disorder (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Antinuclear antibody positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-02-26): https://cdn.clinicaltrials.gov/large-docs/19/NCT03305419/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-30): https://cdn.clinicaltrials.gov/large-docs/19/NCT03305419/SAP_001.pdf